CLINICAL TRIAL: NCT00666601
Title: An Open Label, Single Dose, Microdialysis and Pharmacokinetic Study of TR-701 in Normal Healthy Adults
Brief Title: Microdialysis and Pharmacokinetic Study of TR-701
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1986-022; TR701-102 (Other: TrisuRX Unique ID)
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: Microdialysis; Antibiotic; Healthy subjects
MeSH Terms: interventions — tedizolid; tedizolid phosphate; Prodrugs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilot study (Experimental): 3 subjects, open lable, microdialysis single dose.
  Interventions: Drug: TR-700 (active moiety)
- Main Study (Experimental): 12 subjects, open label, single dose of 600 mg.
  Interventions: Drug: TR-701 (pro-drug)

INTERVENTIONS:
Drug: TR-700 (active moiety) — A TR-700 solution will be locally administered via a microdialysis probe into the skeletal muscle and subcutanous tissue (just under the skin) at a concentration of approximately 2 µg/mL at a flow rate of 1.5 µL/min for 60 minutes for a total maximum dose of 0.36 µg (0.18 µg per probe).
  Arms: Pilot study
Drug: TR-701 (pro-drug) — Each subject enrolled in the Main study will receive a single oral dose of 600mg TR-701
  Arms: Main Study

SUMMARY:
The purpose of this study is to measure the penetration of TR-700 into subcutaneous adipose tissue and skeletal muscle after a single oral dose of 600 mg TR-701

DETAILED DESCRIPTION:
This study will be conducted in two parts: a Pilot Study and a Main Study. The Pilot Study will be conducted to assess recovery of exogenously administered TR-700 (microbiologically active moiety) via microdialysis. In the Main Study, pharmacokinetics of TR-700 will be determined in both soft tissues (via microdialysis) and plasma after a single oral dose of 600 mg TR-701 (prodrug).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 20 to 29 kg/m2
* Agree not to consume any products containing tobacco, alcohol, quinine, grapefruit, caffeine, or high levels of tyramine
* Agree not to use any other medication
* Female subjects must be postmenopausal (for at least 6 months), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control

Exclusion Criteria:

* History of gastric or duodenal ulcer within 1 year before enrollment
* Has known or suspected hypersensitivity or intolerance to heparin, if an indwelling cannula (e.g., heparin lock) is used
* Recent febrile illness (less than 72 hours before the first intake of study medication).
* Significant blood loss (300 mL) or donation of blood within the 60 days before the Screening visit
* Women who are pregnant or breast-feeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04-04 (Actual); Primary Completion 2008-08-12 (Actual); Study Completion 2008-08-12 (Actual)

PRIMARY OUTCOMES:
Subcutaneous tissue concentrations of TR-700 | Single day

CONTACTS AND LOCATIONS:
Overall Officials: Harmut Derendorf, PhD, Principal Investigator — University of Florida
Locations (1):
- General Clinical Research Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sahre M, Sabarinath S, Grant M, Seubert C, Deanda C, Prokocimer P, Derendorf H. Skin and soft tissue concentrations of tedizolid (formerly torezolid), a novel oxazolidinone, following a single oral dose in healthy volunteers. Int J Antimicrob Agents. 2012 Jul;40(1):51-4. doi: 10.1016/j.ijantimicag.2012.03.006. Epub 2012 May 13. PMID 22584101